CLINICAL TRIAL: NCT03269331
Title: Feasibility and Effectiveness of the Advancing Research and Clinical Practice Through Close Collaboration (ARCC) Model for Military Treatment Facility (MTF) Implementation of Nursing Evidence-Based Practice (EBP)
Brief Title: Feasibility and Effectiveness of the Advancing Research and Clinical Practice Through Close Collaboration (ARCC)
Acronym: ARCC
Status: Completed | Type: Observational
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Collaborators: Ohio State University (Other)
Responsible Party: Principal Investigator, Laurie Migliore, Nurse Scientist/Chief, Nursing Research, David Grant U.S. Air Force Medical Center
Other Study IDs: FDG#20160029E
Record Dates: First submitted 2017-08-22; First posted 2017-08-31 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Evidence-Based Practice; Nurse's Role
Keywords: nursing practice; evidence-based practice models; military nursing; clinical inquiry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ARCC EBP Model: CTEP EBP Immersion Course
  Interventions: Behavioral: CTEP EBP Immersion
- Control Group: No CTEP EBP Immersion Course

INTERVENTIONS:
Behavioral: CTEP EBP Immersion — 36 continuing ed credits, virtual library access, collaboration with expert mentors
  Groups: ARCC EBP Model

SUMMARY:
The Institute of Medicine's (IOM) ambitious goal for at least 90% of clinical decisions to be evidence-based includes nursing interventions and practice. Models and frameworks have been developed to meet the demand for practice transformation. While magnet facilities require a commitment to evidence-based nursing practice, military facilities currently lack such a requirement but are instituting evidence-based practice (EBP) initiatives in a purposeful path toward developing high-reliability organizations. Currently, little is known regarding the effectiveness of specific EBP models and frameworks within the military culture. The purpose of this investigation is to determine the effectiveness of the Advancing Research and Clinical Practice through Close Collaboration (ARCC) model in an Air Force Medical Treatment Facility (MTF) beginning with nursing services.

Research questions:

1. What is the current state of organizational culture and readiness for EBP within the MTF's nursing services?
2. Will utilization of the ARCC model significantly improve EBP beliefs, knowledge, and practice in MTF nurses over a two-year period?
3. Is the ARCC model feasible for implementation in Air Force MTF's?

This study includes an intervention group (n=70) of active duty nurses and technicians who attend an intensive 5-day EBP Immersion Workshop and a control group (n=70) who do not. The intervention group will have access to specialized resources such as: a) Center for Transdisciplinary Evidence-Based Practice (CTEP) expert EBP mentors, b) EBP toolkit and resources, c) one year of free access to the Ohio State University (OSU) virtual library. Control group participants will have standard MTF education opportunities. Established valid and reliable survey measures (EBP attitudes, knowledge, beliefs) will be hosted electronically by CTEP at baseline, three, and twelve months. Online measures include institutional and nursing process measures (EBP implementation, policy changes, and publications) over the two-year study period. De-identified data from the anonymous survey measures will be shared by CTEP with this study team. Data analysis will include Student's t-tests to explore differences between groups. Repeated measures ANOVA or the nonparametric equivalent (Friedman's test or Skillings-Mack test) will be used to compare three time points within groups. Feasibility metrics and demographics will be reported with descriptive statistics.

DETAILED DESCRIPTION:
Further study details as provided by David Grant Medical Center, Travis Air Force Base, California

ELIGIBILITY:
Inclusion Criteria:

* Nurse (active duty) assigned to DGMC
* Medical/Surgical technician (active duty) assigned to DGMC
* 15 month retain-ability from time of enrollment

Exclusion Criteria:

* Disciplines outside of Nursing (PA, MD, Occupational Therapy (OT), Physical Therapy (PT), etc.)
* Nurse/technician General Schedule (GS),VA, Contractor employed at David Grant Medical Center (DGMC)
* Anticipated/Scheduled Permanent Change of Station (PCS) in next 15 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: David Grant Medical Center active duty nurses and technicians
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Organizational Culture & Readiness for System-Wide Implementation of EBP Scale (OCRSIEP) changes over time | baseline, month 3, month 12
  25-item assessment of organizational readiness and perceived strengths and barriers for EBP implementation. A 5-point Likert scale with, 1 (not at all) through 5 (very much) measures item response to questions focused on the extent that EBP is included in current organizational culture. For example, "To what extend do you believe that EBP is practiced in your organization?" Overall, the instrument measures the relationship between cultural factors and the organization's implementation of EBP over a 6-month time frame. Validity is reported with content and face validity and internal consistency reliabilities greater than 0.85
Evidence-Based Practice Beliefs (EBPB) Scale changes over time | baseline, month 3, month 12
  16-item assessment of an individual's beliefs regarding the value of EBP and capability for EBP implementation in clinical nursing practice. A 5-point Likert scale with, 1 (strongly disagree) through 5 (strongly agree) measures item response to statements about EBP, such as: "I believe EBP takes too much time"… "I am clear about the steps of EBP." It is anticipated, based on the results of several studies, that higher scores on the EBPB scale are associated with greater implementation of EBP and better healthcare outcomes. Validity is reported with content and face validity as well as internal consistency reliabilities greater than 0.85.
Evidence-Based Practice Implementation (EBPI) Scale changes over time | baseline, month 3, month 12
  18-item instrument to measure the extent to which healthcare workers integrate scientific evidence in their clinical practice. A 5-point ordinal scale with frequencies listed from 0 times (0 pt.), 1-3 times (1 pt.), 4-5 times (2 pt.), 6-7 times (3 pt.) and > 8 times (4 pt.) is used to assess how often each item has applied over the past 8 weeks. For example, how often have you: "Used evidence to change my clinical practice…", "Accessed the National Guidelines Clearinghouse…" Total scores are summed where higher scores indicate greater integration of EBP in the healthcare workers practice. Validity is reported with content and face validity as well as internal consistency reliabilities greater than 0.85.
EBP Knowledge Assessment Questionnaire (EBP-KAQ) changes over time | baseline, month 3, month 12
  27-item multiple-choice objective knowledge measure of examine EBP knowledge.

SECONDARY OUTCOMES:
Nursing process outcomes changes over time | baseline, month 3, month 12
  projects, policy changes, publications

OTHER OUTCOMES:
Feasibility metrics changes over time | baseline, month 3, month 12
  Costs, mentors, staff retention

CONTACTS AND LOCATIONS:
Overall Officials: Laurie A Migliore, PhD, Principal Investigator — Staff
Locations (1):
- David Grant Medical Center, Fairfield, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Breckenridge-Sproat ST, Throop MD, Raju D, Murphy DA, Loan LA, Patrician PA. Building a Unit-Level Mentored Program to Sustain a Culture of Inquiry for Evidence-Based Practice. Clin Nurse Spec. 2015 Nov-Dec;29(6):329-37. doi: 10.1097/NUR.0000000000000161. PMID 26444511
- [Background] Barrera M Jr, Castro FG, Strycker LA, Toobert DJ. Cultural adaptations of behavioral health interventions: a progress report. J Consult Clin Psychol. 2013 Apr;81(2):196-205. doi: 10.1037/a0027085. Epub 2012 Jan 30. PMID 22289132
- [Background] Bryan CJ, Jennings KW, Jobes DA, Bradley JC. Understanding and preventing military suicide. Arch Suicide Res. 2012;16(2):95-110. doi: 10.1080/13811118.2012.667321. PMID 22551041
- [Background] Committee on the Assessment of Resiliency and Prevention Programs for Mental and Behavioral Health in Service Members and Their Families; Board on the Health of Select Populations; Institute of Medicine; Denning LA, Meisnere M, Warner KE, editors. Preventing Psychological Disorders in Service Members and Their Families: An Assessment of Programs. Washington (DC): National Academies Press (US); 2014 Feb 11. Available from http://www.ncbi.nlm.nih.gov/books/NBK222170/ PMID 25057692
- [Background] Kenny DJ, Richard ML, Ceniceros X, Blaize K. Collaborating across services to advance evidence-based nursing practice. Nurs Res. 2010 Jan-Feb;59(1 Suppl):S11-21. doi: 10.1097/NNR.0b013e3181c3c011. PMID 20010273
- [Background] Melnyk BM. Achieving a high-reliability organization through implementation of the ARCC model for systemwide sustainability of evidence-based practice. Nurs Adm Q. 2012 Apr-Jun;36(2):127-35. doi: 10.1097/NAQ.0b013e318249fb6a. PMID 22407205
- [Background] Melnyk BM, Bullock T, McGrath J, Jacobson D, Kelly S, Baba L. Translating the evidence-based NICU COPE program for parents of premature infants into clinical practice: impact on nurses' evidence-based practice and lessons learned. J Perinat Neonatal Nurs. 2010 Jan-Mar;24(1):74-80. doi: 10.1097/JPN.0b013e3181ce314b. PMID 20147834
- [Background] Melnyk BM, Fineout-Overholt E, Giggleman M, Cruz R. Correlates among cognitive beliefs, EBP implementation, organizational culture, cohesion and job satisfaction in evidence-based practice mentors from a community hospital system. Nurs Outlook. 2010 Nov-Dec;58(6):301-8. doi: 10.1016/j.outlook.2010.06.002. PMID 21074647
- [Background] Melnyk BM, Fineout-Overholt E, Gallagher-Ford L, Kaplan L. The state of evidence-based practice in US nurses: critical implications for nurse leaders and educators. J Nurs Adm. 2012 Sep;42(9):410-7. doi: 10.1097/NNA.0b013e3182664e0a. PMID 22922750
- [Background] Melnyk BM, Gallagher-Ford L, Thomas BK, Troseth M, Wyngarden K, Szalacha L. A Study of Chief Nurse Executives Indicates Low Prioritization of Evidence-Based Practice and Shortcomings in Hospital Performance Metrics Across the United States. Worldviews Evid Based Nurs. 2016 Feb;13(1):6-14. doi: 10.1111/wvn.12133. Epub 2016 Feb 1. PMID 26873371
- [Background] Muller A, McCauley K, Harrington P, Jablonski J, Strauss R. Evidence-based practice implementation strategy: the central role of the clinical nurse specialist. Nurs Adm Q. 2011 Apr-Jun;35(2):140-51. doi: 10.1097/NAQ.0b013e31820f47e9. PMID 21403488
- [Background] Sackett DL, Rosenberg WM, Gray JA, Haynes RB, Richardson WS. Evidence based medicine: what it is and what it isn't. BMJ. 1996 Jan 13;312(7023):71-2. doi: 10.1136/bmj.312.7023.71. No abstract available. PMID 8555924
- [Background] Sammer CE, Lykens K, Singh KP, Mains DA, Lackan NA. What is patient safety culture? A review of the literature. J Nurs Scholarsh. 2010 Jun;42(2):156-65. doi: 10.1111/j.1547-5069.2009.01330.x. PMID 20618600
- [Background] Ubbink DT, Guyatt GH, Vermeulen H. Framework of policy recommendations for implementation of evidence-based practice: a systematic scoping review. BMJ Open. 2013 Jan 24;3(1):e001881. doi: 10.1136/bmjopen-2012-001881. PMID 23355664
- [Background] Wallen GR, Mitchell SA, Melnyk B, Fineout-Overholt E, Miller-Davis C, Yates J, Hastings C. Implementing evidence-based practice: effectiveness of a structured multifaceted mentorship programme. J Adv Nurs. 2010 Dec;66(12):2761-71. doi: 10.1111/j.1365-2648.2010.05442.x. Epub 2010 Sep 6. PMID 20825512
- [Background] Williamson KM, Almaskari M, Lester Z, Maguire D. Utilization of evidence-based practice knowledge, attitude, and skill of clinical nurses in the planning of professional development programming. J Nurses Prof Dev. 2015 Mar-Apr;31(2):73-80. doi: 10.1097/NND.0000000000000140. PMID 25790357
- [Background] Wilson M, Sleutel M, Newcomb P, Behan D, Walsh J, Wells JN, Baldwin KM. Empowering nurses with evidence-based practice environments: surveying Magnet(R), Pathway to Excellence(R), and non-magnet facilities in one healthcare system. Worldviews Evid Based Nurs. 2015 Feb;12(1):12-21. doi: 10.1111/wvn.12077. Epub 2015 Jan 16. PMID 25598144